CLINICAL TRIAL: NCT06510569
Title: Three-Dimensional Evaluation of Clear Aligners Versus Fixed Orthodontic Treatment of Lower Anterior Crowding: A Randomized Clinical Trial
Brief Title: 3D Evaluation of Clear Aligners Versus Fixed Orthodontic Treatment of Lower Anterior Crowding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haidy Fekry (Other Government)
Responsible Party: Sponsor-Investigator, Haidy Fekry, dentist, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-I
Record Dates: First submitted 2024-06-20; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pathological Resorption of External Root

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear aligner therapy (Experimental): U lab aligners
  Interventions: Device: U lab aligners
- Fixed orthodontic treatment (Experimental): Oromo bracket
  Interventions: Device: oramco bracket

INTERVENTIONS:
Device: U lab aligners — Aligner group change the aligner every 10 days
  Arms: Clear aligner therapy
Device: oramco bracket — changing orthodontic wire every one month
  Arms: Fixed orthodontic treatment

SUMMARY:
Evaluate and compare clear aligners versus fixed orthodontic treatment of lower anterior crowding with the use of cone-beam computed tomography within maximum 6 months or until correction of lower anterior crowding whichever is nearest to occur.

DETAILED DESCRIPTION:
Group (A): Patients will be treated with conventional fixed orthodontic treatment in lower anterior crowding.

Group (B): Patients will be treated with clear aligner therapy in lower anterior crowding.

ELIGIBILITY:
Inclusion Criteria:

Adult female patients . age 18-25 y . Patients with mild to moderate lower anterior crowding (1 mm - 6 mm ) . Healthy compliant and motivated patient . full dentition except wisdom teeth .

Exclusion Criteria:

Previous orthodontic treatments. Any systemic disease Pregnant and lactating female. pocket depth more than 5 mm.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Correction of lower anterior crowding | 6 months
  according to little irregularity index

OTHER OUTCOMES:
Root resorption | 6 month
  CBCT evaluation of root resorption

CONTACTS AND LOCATIONS:
Overall Officials: samir A ibrahim, proffesor, Principal Investigator — Al azhar universty
Locations (2):
- Egypt (2):
  - Al Azhar Universty, Cairo
  - Haidy Fekry, Zagazig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fiori A, Minervini G, Nucci L, d'Apuzzo F, Perillo L, Grassia V. Predictability of crowding resolution in clear aligner treatment. Prog Orthod. 2022 Nov 28;23(1):43. doi: 10.1186/s40510-022-00438-z. PMID 36437397
- See also: Predictability of crowding resolution in clear aligner treatment — https://pubmed.ncbi.nlm.nih.gov/36437397/

DOCUMENTS (1):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT06510569/Prot_000.pdf